CLINICAL TRIAL: NCT01030224
Title: A Phase-1, Single Center, Double Blind, Randomized, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Intravenous AZD9742 After Single Ascending Doses in Healthy Male and Female Subjects
Brief Title: This is a Study to Evaluate the Safety, Tolerability and Pharmacokinetics (PK) of AZD9742 After Single IV Doses in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D2690C00001
Record Dates: First submitted 2009-12-09; First posted 2009-12-11 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: Healthy volunteer; First time in human

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AZD9742 IV Infusion (Experimental): Active
  Interventions: Drug: AZD9742
- Placebo to AZD9742 IV Infusion (Placebo Comparator): Placebo
  Interventions: Drug: Placebo to match AZD9742

INTERVENTIONS:
Drug: AZD9742 — Increasing single IV infusion doses of AZD9742 given to approximately 6 cohorts of 8 subjects each (6 on active and 2 on placebo). Specific doses will be selected by the safety review committee
  Arms: AZD9742 IV Infusion
Drug: Placebo to match AZD9742 — Single IV infusion of AZD9742 placebo given to approximately 6 cohorts of 8 subjects each (6 on active and 2 on placebo)
  Arms: Placebo to AZD9742 IV Infusion

SUMMARY:
The main purpose of this study is to assess the safety, tolerability and PK of AZD9742 after single IV doses.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Clinically normal physical findings and laboratory values as judged by the investigator with normal ECG.
* Healthy male and female volunteers. Females must be of non childbearing potential.

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within 4 weeks of the first administration of the Investigational Product
* History of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AZD9742 will be assessed by incidence and severity of AE's, abnormalities in vital signs, ECG's, telemetry, clinical laboratory assessments, physical exams and withdrawals | Assessments taken at Visit 1 (enrollment), defined timepoints pre-dose and post-dose during Visit 2 (residential period) and at Visit 3 (follow up). Volunteers will be monitored througout the study from Visit 1 through Visit 3 for adverse events.

SECONDARY OUTCOMES:
Pharmacokinetic profile: to characterize the pharmacokinetics of AZD9742 in blood and urine | Samples taken during Visit 2 (residential period) at defined timepoints pre-dose and post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ralph A Schutz, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States